CLINICAL TRIAL: NCT05947318
Title: Effect of Transcranial Alternating Current Stimulation on the Recovery of Motor Control of the Upper Limb and Cerebral Connectivity in Chronic-stage Stroke Patients
Brief Title: Effect of tACS on the Recovery of Motor Control of the Upper Limb and Cerebral Connectivity in Chronic Stroke Patients
Acronym: tACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Metropolitana de Ciencias de la Educacion (Other)
Responsible Party: Principal Investigator, Juan Jose Mariman Rivero, Full professor, Universidad Metropolitana de Ciencias de la Educacion
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: FONDECYT N° 11221226
Record Dates: First submitted 2023-06-12; First posted 2023-07-17 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Chronic Stroke; Rehabilitation
Keywords: transcranial alternating current stimulation; motor recovery; stroke rehabilitation

STUDY DESIGN:
Intervention Model Description: Three experimental groups:
  1. tACS-70 Hz group
  2. tACS-7Hz group
  3. tACS-sham group
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Neither the participant or the professionals that will make the training and the assessments will know to which group the participants was assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- tACS - 70 Hz group (Experimental): The group will receive the training program plus 20 minutes of tACS at 70 Hz in the C3 or C4 electrode position (depending of the hemiparetic arm) during a specific kinetic and kinematic tasks in every training session.
  Interventions: Device: transcranial alternating current stimulation 70 Hz; Behavioral: Training
- tACS - 7 Hz group (Active Comparator): The group will receive the training program plus 20 minutes of tACS at 7 Hz in the C3 or C4 electrode position (depending of the hemiparetic arm) during a specific kinetic and kinematic tasks in every training session.
  Interventions: Behavioral: Training; Device: transcranial alternating current stimulation 7 Hz
- tACS - sham group (Sham Comparator): The group will receive the training program plus 30 seconds of tACS at 70 Hz in the C3 or C4 electrode position (depending of the hemiparetic arm) in every training session.
  Interventions: Behavioral: Training; Device: transcranial alternating current stimulation Sham

INTERVENTIONS:
Device: transcranial alternating current stimulation 70 Hz — Transcranial alternating current stimulation in the head above the motor cortex area of one side of the brain, according to the hemiparesis side.
  Electrodes with 3.14 cm2 of stimulation area will be used, therefore, the initial current intensity will be 0.21 mA, with a current density of 0.07 mA / cm2. The current intensity will be adjusted to the tactile sensory threshold and phosphenes of each patient, with in order to reduce such sensory effects, but considering that the decrease in current will not be greater than 10% of the initial intensity, in order to obtain a comparable configuration between subjects.
  The frequency stimulation will be 70 Hz
  Arms: tACS - 70 Hz group
Behavioral: Training — Training of the upper limb with specific kinematic and kinetic tasks plus functional training
Device: transcranial alternating current stimulation 7 Hz — Transcranial alternating current stimulation in the head above the motor cortex area of one side of the brain, according to the hemiparesis side.
  Electrodes with 3.14 cm2 of stimulation area will be used, therefore, the initial current intensity will be 0.21 mA, with a current density of 0.07 mA / cm2. The current intensity will be adjusted to the tactile sensory threshold and phosphenes of each patient, with in order to reduce such sensory effects, but considering that the decrease in current will not be greater than 10% of the initial intensity, in order to obtain a comparable configuration between subjects.
  The frequency stimulation will be 7 Hz
  Arms: tACS - 7 Hz group
Device: transcranial alternating current stimulation Sham — Transcranial alternating current stimulation in the head above the motor cortex area of one side of the brain, according to the hemiparesis side.
  Electrodes with 3.14 cm2 of stimulation area will be used, therefore, the initial current intensity will be 0.21 mA, with a current density of 0.07 mA / cm2. The current intensity will be adjusted to the tactile sensory threshold and phosphenes of each patient, with in order to reduce such sensory effects, but considering that the decrease in current will not be greater than 10% of the initial intensity, in order to obtain a comparable configuration between subjects.
  The stimulation will be turn on for 30 seconds (at 70 Hz)
  Arms: tACS - sham group

SUMMARY:
This project seeks to evaluate the effect of transcranial alternating current stimulation (tACS) on the recovery of motor control of the upper limb and associated neuronal synchrony during a 14-sessions (5-week) rehabilitation program for adult patients with diagnosis of stroke at chronic stage. Specifically, the stimulation on Gamma ranges, because the evidence available so far allows us to propose that the tACS in the Gamma range (around 70 Hz) facilitates motor execution.

For this purpose, the experimental approach involves active (70 Hz in Gamma rhythm and 7 Hz, Theta rhythm) and sham tACS together with an analytical and integrated motor training with a double-blind and randomized design.

Our hypothesis is that Gamma frequency tACS restores neuronal synchrony in Beta range, which enhances the upper limb motor recovery associated with a training program.

Using specific motor control parameters, clinical scales and electroencephalography, the immediate and long-term (3 months after finished the training) behavioral and neurophysiological effect of this new neurostimulation paradigm (tACS plus training) for motor rehabilitation of stroke will be established.

DETAILED DESCRIPTION:
This project seeks to evaluate the effect of transcranial alternating current stimulation (tACS) on the recovery of motor control of the upper limb and associated neuronal synchrony during a 14 sessions (5 week) rehabilitation program for adult patients with diagnosis of stroke at chronic stage. Specifically, the stimulation on Gamma ranges, because the evidence available so far allows us to propose that the tACS in the Gamma range (around 70 Hz) facilitates motor execution. For this purpose, the experimental approach involves active (70 Hz in Gamma rhythm and 7 Hz, Theta rhythm) and sham tACS together with an analytical and integrated motor training with a double-blind and randomized design.

Our hypothesis is that Gamma frequency tACS restores neuronal synchrony in Beta range, which enhances the upper limb motor recovery associated with a training program.

The general objective is to assess the effects of a combined program of tACS and upper limb training on motor performance and brain connectivity in chronic-stage stroke patients.

The specifics objectives to accomplish this are (1) Implement a system for simultaneous measurement of motor activity and EEG under tACS, considering possible postural alterations in stroke patients. (2) Evaluate the upper limb motor control and neuronal synchrony associated with motor performance during the execution of a combined stimulation and training program. Training will include analytical and functional tasks to optimize the performance in function and activity ICF level. tACS will be applied only during analytical task. (3) Analyze the changes in motor performance and neuronal synchrony for the experimental groups.

Using specific motor control parameters (kinetic and kinematic control), clinical scales and electroencephalography, the immediate and long-term (3 months after finished the training) behavioral and neurophysiological effect of this new neurostimulation paradigm (tACS plus training) for motor rehabilitation of stroke will be established.

By means of analysis of variance, clustering comparisons and linear regressions, it will be established the effect of tACS on neuronal synchrony and the parallel motor activity, as well as their underlying relationship.

We will use the REDCap platform to register all the clinical data given by the medical record and clinical assessments.

The recruitment will be made at the Clinical Center of Metropolitan University of Educational Sciences and in the Primary Care Centers that are near to the University. The sample size is 45 chronic stage stroke survivors. The sample size calculation used the data available in the study for the difference in Fugl-Meyer score between the bihemispheric and sham transcranial Direct Current Stimulation groups after the intervention (in the study of Alisar et al, 2020), considering an effect size of 1.4, a p-value of 0.05 and a power (1- beta) of 0.9, which yielded a sample size of 12 subjects per group. Now, also considering an attrition percentage of 20% and an equivalence in the size of the 3 study groups, the final sample size is 15 people per group (45 people in total).

To answer the study hypothesis, two variables will be examined as primary results:

1. Behavioral level, it will be the score on the Fugl-Meyer scale (upper extremity section). This scale has been widely used in the field of neurorehabilitation to assess motor impairments (ICF function level).
2. Neurophysiological level, the primary outcome will be the change in spectral power in the Beta band (13-30Hz) associated with motor performance in kinetic and kinematic tasks. Signal processing will follow a cluster approach using the Fieldtrip toolbox in Matlab software (R2016B).

Both variables will be subjected to a two-factor analysis of variance (experimental group factor (3 levels, tACS-70Hz, 7Hz and simulated) and time factor (4 levels referred to the measurement times)). Depending on the result, it will apply a post-hoc test (bonferroni) to study differences between levels and interactions. The association between the variables will be inspected through regression models. The level of significance will have a p-value of 0.05. The statistical analysis will be implemented in the R language and the Rstudio software. Complementary to the primary results, and in order to broaden the description of the study phenomenon, the scores of the clinical scales already described will be analyzed, as well as kinetic (absolute force, speed of force change) and kinematic variables (direction error, maximum speed) of the analytical and combined tasks. In addition, the long-scale synchrony will be described by means of connectivity variables between the electrodes already identified (phase locking value and weighted phase lag index).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unilateral stroke at chronic stage (6 months or more)
* Upper Extremity -Fugl Meyer > 10
* Wrist extensors strength of the paretic limb of 2 or more in the Medical Research Council (MRC) scale
* Active shoulder movement (flexion or abduction) of 30º or more
* Be able to follow the instructions necessary to achieve the training protocol

Exclusion Criteria:

* Have a cerebellar stroke or ataxia
* Have some medical condition contraindicated for tACS (epilepsy, pacemaker, prosthesis between others)
* Have post-stroke epilepsy
* Limited passive range of motion in the elbow (less than 45º in flexo-extension plane)
* Limited passive range of motion in the wrist (less than 40º in flexo-extension plane)
* Limited passive range of motion in the shoulder (less than 70º in flexo-extension plane)
* Have another neurological condition that leads to upper extremity sequelae
* Have a normal performance in the clinical test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Impairment Measure pre-intervention: Upper Extremity Fugl Meyer | week 0
  Scale use to assess motor impairments (ICF function level), and adequately reflects the analytical motor control of force and direction of movement. The scale has a maximum of 66 points, which indicates a normal performance. Lower scores indicate worse performance.
Change of Impairment Measure post-intervention: Upper Extremity Fugl Meyer | week 5 or 6 (end of the training program)
  Scale use to assess motor impairments (ICF function level), and adequately reflects the analytical motor control of force and direction of movement. The scale has a maximum of 66 points, which indicates a normal performance. Lower scores indicate worse performance.
Change of Impairment Measure follow up: Upper Extremity Fugl Meyer | week 12
  Scale use to assess motor impairments (ICF function level), and adequately reflects the analytical motor control of force and direction of movement. The scale has a maximum of 66 points, which indicates a normal performance. Lower scores indicate worse performance.
EEG spectral power in Beta band pre-intervention | week 0
  Change in spectral power in the Beta band (13-30Hz) associated with motor performance in kinetic and kinematic tasks
Change in EEG spectral power in Beta band post-intervention | week 5 or 6 (end of the training program)
  Change in spectral power in the Beta band (13-30Hz) associated with motor performance in kinetic and kinematic tasks
Change in EEG spectral power in Beta band follow up | week 12
  Change in spectral power in the Beta band (13-30Hz) associated with motor performance in kinetic and kinematic tasks

SECONDARY OUTCOMES:
Activity Measure: Action Research Arm Test | week 0, week 5 or 6 (end of the training program) and week 12
  Action Research Arm Test will be used to evaluate de ICF activity level. The maximum score is 57, which indicate a normal perfomance. Lower scores indicate worse performance.
Change in Activity Measure post-intervention: Action Research Arm Test | week 5 or 6 (end of the training program)
  Action Research Arm Test will be used to evaluate de ICF activity level. The maximum score is 57, which indicate a normal perfomance. Lower scores indicate worse performance.
Change in Activity Measure follow up: Action Research Arm Test | week 12
  Action Research Arm Test will be used to evaluate de ICF activity level. The maximum score is 57, which indicate a normal perfomance. Lower scores indicate worse performance.
Performance measure in the trained kinetic task (behavioral parameter) | week 0, week 5 or 6 (end of the training program) and week 12
  The change that we observed in the kinetic task in the protocol training. This outcome is a behavioral parameter that measures the change in the task that is trained in the training protocol. It is a measure of how the participants performed the kinetic task
Change in the performance measure in the trained kinetic task post-intertenvion (behavioral parameter) | week 5 or 6 (end of the training program)
  The change that we observed in the kinetic task in the protocol training. This outcome is a behavioral parameter that measures the change in the task that is trained in the training protocol. It is a measure of the change in the performance in the kinetic task at the beginning of the training protocol and at the end.
Change in the performance measure in the trained kinetic task at follow up (behavioral parameter) | week 12
  The change that we observed in the kinetic task in the protocol training. This outcome is a behavioral parameter that measures the change in the task that is trained in the training protocol. It is a measure of the change in the performance in the kinetic task at the beginning of the training protocol and at the 12 week follow up.
Performance measure in trained kinematic task (behavioral parameter) | week 0, week 5 or 6 (end of the training program) and week 12
  The change that we observed in the kinematic task in the protocol training. This outcome is a behavioral parameter that measures the change in the task that is trained in the training protocol. It is a measure of how the participants performed the kinematic task
Change in the performance measure in the trained kinematic task post-intervention (behavioral parameter) | week 5 or 6 (end of the training program)
  The change that we observed in the kinematic task in the protocol training. This outcome is a behavioral parameter that measure the change in the task that is trained in the training protocol. It is a measure of the change in the performance in the kinematic task at the beginning of the training protocol and at the end.
Change in performance measure in the trained kinematic task at follow up (behavioral parameter) | week 12
  The change that we observed in the kinematic task in the protocol training. This outcome is a behavioral parameter that measure the change in the task that is trained in the training protocol. It is a measure of the change in the performance in the kinematic task at the beginning of the training protocol and at the end.

CONTACTS AND LOCATIONS:
Overall Officials: Juan J Mariman, Ph.D, Principal Investigator — Universidad Metropolitana de Ciencias de la Educacion
Locations (1):
- Centro de Habilidades Clínicas - Universidad Metropolitana de Ciencias de la Educación, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
For now, we have no plans of sharing individual participant data.

REFERENCES:
- [Background] Alisar DC, Ozen S, Sozay S. Effects of Bihemispheric Transcranial Direct Current Stimulation on Upper Extremity Function in Stroke Patients: A randomized Double-Blind Sham-Controlled Study. J Stroke Cerebrovasc Dis. 2020 Jan;29(1):104454. doi: 10.1016/j.jstrokecerebrovasdis.2019.104454. Epub 2019 Nov 4. PMID 31699572